CLINICAL TRIAL: NCT06747559
Title: Effects of Vitamin D Supplementation on Postoperative Rehabilitation in Hip and Knee Osteoarthritis Patients: a Multicenter Randomized Controlled Trial
Brief Title: Effects of Vitamin D Supplementation on Postoperative Rehabilitation in Hip and Knee Osteoarthritis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Yiwu Fuyuan Private Hospital (Unknown); Hangzhou Xiaoshan Traditional Chinese Orthopedic Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-1022
Record Dates: First submitted 2024-11-21; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis of the Hip or Knee; Joint Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D oral supplement (Experimental): Using vitamin D oral supplement that has been widely used in clinic
  Interventions: Drug: Vitamin D
- No vitamin D supplementation (No Intervention)

INTERVENTIONS:
Drug: Vitamin D — Vitamin D oral supplementation
  Arms: Vitamin D oral supplement

SUMMARY:
The goal of this clinical trial is to learn if vitamin D supplementation affects postoperative rehabilitation in osteoarthritis patients who underwent joint arthroplasty. The main questions it aims to answer are:

Does oral vitamin D supplementation for a period of time after joint arthroplasty affect the postoperative recovery speed in patients who have vitamin D deficiency? Does oral vitamin D supplementation after joint arthroplasty affect the long-term recovery of joint functions in patients who have vitamin D deficiency?

Participants will:

Take vitamin D oral supplement every day for 3 months. Visit the clinic in 1, 3, 6, 12 months after joint replacement surgery for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

1. Vitamin D deficiency (blood 25-hydroxyvitamin D value < 20ng/ml);
2. Meeting the diagnostic criteria for hip or knee osteoarthritis;
3. Planning to undergo hip or knee arthroplasty after clinical assessment;

Exclusion Criteria:

1. Having other diseases that could cause damage to the bone or cartilage structure of the hip or knee, such as trauma, joint infection, congenital joint malformation, and systemic diseases such as rheumatoid arthritis and gout.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee joint function | From enrollment to the end of treatment at 1 year
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). Pain ranging from 0 to 20 points; stiffness, 0 to 8 points; and physical function, 0 to 68 points. Higher scores represent worse pain, stiffness, and functional limitations.
Hip joint function | From enrollment to the end of treatment at 1 year
  Harris Hip Score. The maximum score possible is 100. Results can be interpreted with the following: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.
Muscle strength | From enrollment to the end of treatment at 1 year
  Using portable muscle strength tester to measure flexor and extensor muscle strength of knee or hip joint

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Zhao, MD, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
IPD cannot be shared publicly due to the sponsor policy.